CLINICAL TRIAL: NCT01752426
Title: A Pilot Study to Determine the Effects of the Bruton's Tyrosine Kinase (Btk) Inhibitor PCI-32765 on Leukemia Cell Kinetics and Trafficking, Using Heavy Water Labeling in Subjects With Chronic Lymphocytic Leukemia (CLL) and Small Lymphocytic Lymphoma (SLL)
Brief Title: Pilot Study to Determine Effects of the Btk Inhibitor PCI-32765 on Leukemia Cell Kinetics and Trafficking, Using Heavy Water Labeling in Subjects With CLL and SLL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0086; NCI-2013-00029 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-12-13; First posted 2012-12-19 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Leukemia
Keywords: Leukemia; Chronic Lymphocytic Leukemia; CLL; Small Lymphocytic Lymphoma; SLL; PCI-32765; Ibrutinib; Btk inhibitor; Heavy water; 2H2O
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Deuterium Oxide; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Heavy Water + PCI-32765 (Experimental): Subjects given 50ml 70% 2H2O (Heavy Water) 3 times a day for the first 5 days followed by 60 ml daily for a total of 4 weeks (labeling phase). Subjects given first dose in clinic. Subjects then given individual doses of 2H2O to consume at home; after the 5-day loading period, a 60 ml maintenance dose of 2H2O will be drunk at bedtime. At end of the 4th week, subjects stop drinking 2H2O (washout phase) and be followed from 6-12 weeks until beginning treatment with PCI-32765. PCI-32765 administered with 8 ounces (~240mL) of water at a dose of 420 mg (3 x 140mg capsules) orally once daily and continued daily. Treatment duration is 12 cycles, with each cycle consisting of 28 days.
  Interventions: Other: Heavy Water (2H2O); Drug: PCI-32765

INTERVENTIONS:
Other: Heavy Water (2H2O) — 50 ml 70% 2H2O 3 times a day for the first 5 days followed by 60 ml daily for a total of 4 weeks. After the 5-day loading period, a 60 ml maintenance dose of 2H2O will be drunk at bedtime. At end of the 4th week, subjects stop drinking 2H2O (washout phase) and be followed from 6-12 weeks until beginning treatment with PCI-32765.
Drug: PCI-32765 — 420 mg orally once daily.
  Other Names: Ibrutinib

SUMMARY:
The goal of this clinical research study is to learn how PCI-32765 (ibrutinib) may affect the life cycle of blood-cancer cells. Cancer cells will be "labeled" with heavy water to learn about their birth rates and death rates.

Ibrutinib is a type of drug called a kinase inhibitor. Kinases are proteins inside cells that help cells live and grow. The study drug is designed to inhibit or "block" the activity of a type of kinase that helps blood-cancer cells live and grow. By blocking the activity of this specific kinase, it is possible that the study drug may kill the cancer cells or stop them from growing.

Heavy water (2H2O) is a special type of water that is designed to help researchers learn how quickly cancer cells in the body reproduce.

DETAILED DESCRIPTION:
Heavy Water Administration:

If you are found to be eligible to take part in this study, you will receive heavy water to drink for 4 weeks. The vials of heavy water will be shipped to your home location.

On Days 1-5, you will drink the heavy water 3 times each day. You will drink 1 dose in the morning, 1 dose in the afternoon, and 1 dose in the evening. You should take the doses at least 3 hours apart. If you miss a dose, take it as soon as you remember. Make sure to wait at least 3 hours between doses.

Starting on Day 6 and until your first study visit, you will drink the heavy water 1 time each day in the evening.

You may choose to drink the heavy water with or without food.

You will be given a study diary to record your doses. If you miss a dose, take it as soon as you remember. If you vomit a dose, you do not need to make it up. Just wait until the next regularly scheduled dose and make a note of it in the diary.

Heavy Water Study Visits:

On Day 1 and during Weeks 2 and 4, blood (about 5 tablespoons) will be drawn for routine tests and for heavy water testing. These blood samples will not be banked for future research. The samples will only be used for research in this study and will be kept until all DNA and protein analysis is complete. These Samples will be sent to our collaborators at the Feinstein Institute for Medical Research and KineMed, Inc., in order to conduct the heavy water analyses.

After Week 4, you will stop drinking the heavy water and will be followed either in the clinic or by your local doctor for 6-12 weeks.

Every 2 weeks during the time after you stop drinking heavy water and before you start taking ibrutinib, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* Blood (about 4 tablespoons) will be drawn for heavy water testing. This measures how fast the cancer cells are making new protein and DNA.
* You will be asked about any drugs you may be taking.

Every 4 weeks during the time after you stop drinking heavy water and before you start taking ibrutinib, blood (about 1 tablespoon) will be drawn for routine tests.

Ibrutinib Administration:

Beginning around Weeks 10-16, you will start taking ibrutinib. You will take 3 capsules by mouth with 1 cup (8 ounces) of water 1 time a day. The dose should be taken at least 30 minutes before eating and at least 2 hours after a meal, at about the same time each day.

If you miss or vomit a dose, do not make up the dose. Take the next dose at your regularly scheduled time and be sure to write it down in the study diary.

You will take the study drug for up to 12 cycles. Each cycle is 28 days. If the doctor thinks it is in your best interest, you may continue taking the study drug even after 12 cycles.

You will also take allopurinol by mouth 1 time each day during the first 1-2 weeks of taking ibrutinib to lower the risk of side effects.

Ibrutinib Study Visits:

At every study visit, you will be asked about any drugs you may be taking and about any side effects you may be having.

On Days 1 and 3 of Week 1, and at the end of Weeks 2, 4, 6, 8, and 10:

* You will have a physical exam, including measurement of your vital signs.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* Blood (about 4 tablespoons) will be drawn for heavy water testing.

At the end of Week 12:

* You will have a physical exam, including measurement of your vital signs.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* Blood (about 4 tablespoons) will be drawn for heavy water testing.
* You will have computed tomography (CT) scans of the chest, abdomen, and pelvis to check the status of the disease.
* You will have a bone marrow aspiration to check the status of the disease. To collect a bone marrow aspirate, an area of the hip or other site is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle.

At the end of Weeks 16 and 20:

* You will have a physical exam, including measurement of your vital signs.
* Blood (about 2 tablespoon) will be drawn for routine tests.

At the end of Weeks 24 and 36:

* You will have a physical exam, including measurement of your vital signs.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will have CT scans to check the status of the disease.
* You will have a bone marrow aspiration to check the status of the disease.

At the end of Week 48:

* You will have a physical exam, including measurement of your vital signs.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will have CT scans to check the status of the disease.

Length of Study Drug Dosing:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the end-of-study visits.

Follow-Up Visi:

If you continue taking the study drug past 12 cycles, you will come to the clinic for follow-up visits every month. You will continue to have follow-up visits as long as you are taking the study drug. At each visit, the following tests and procedures will be performed:

You will have a physical exam, including measurement of you vital signs. Blood (about 1 tablespoon) will be drawn for routine tests.

Whenever the doctor thinks it is needed, you will have the following tests and procedures:

You may have CT scans to check the status of the disease. You may have a bone marrow aspiration to check the status of the disease.

End-of-Study Visits:

After your last dose of study drug, and then 1 more time during the next month, you will have end-of-study visits. The following tests and procedures will be performed:

You will have a physical exam, including measurement of you vital signs. You will be asked about any symptoms you may be having. Blood (about 1 tablespoon) will be drawn for routine tests.

This is an investigational study. Ibrutinib is FDA approved and commercially available for the treatment of patients with mantle cell lymphoma. Its use in this study is investigational.

Up to 30 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of CLL/ SLL and have not been previously treated.
2. An indication for treatment by 2008 IWCLL Criteria.
3. Male and female subjects of age >/= 18 years at the time of signing informed consent and requiring treatment within the next 2 to 6 months.
4. Understand and voluntarily sign an informed consent, and be able to comply with study procedures and follow-up examinations.
5. Platelet counts at study entry must be greater than 50,000/µL and absolute neutrophil counts at study entry must be greater than 750/µL.
6. Free of prior malignancies for 3 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix or breast.
7. Subjects must be able to contribute the required amount of blood and/or tissue without compromising their well-being or care and must weigh at least 110 pounds.
8. Adequate renal and hepatic function as indicated by all of the following: total bilirubin </=1.5 x institutional Upper Limit of Normal (ULN); Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) </=2.5 x Upper limits of normal (ULN); and estimated creatinine clearance (CrCl) of > 30 mL/min, as calculated by the Cockcroft-Gault equation.
9. Participants must be willing to be contacted again for consideration of additional studies in the future, such as a blood draw or another action (e.g., bone marrow aspiration and/or biopsy) that would be associated with their standard of care, unless they consented to such for research purposes.
10. An Eastern Cooperative Oncology (ECOG)/World Health Organization (WHO) performance status of 0-2.
11. Males and females of child bearing potential must have adequate birth control protection while on study and for 30 days after the last dose of study drug. The couple will use two forms of birth control for the entire time of the study and 30 days after finishing study. Conception control should include a hormonal method (birth control pill, etc.), and a double-barrier methods (condoms with spermicidal, sponge with spermicidal, or diaphragm with spermicidal), or abstinence (not having sex) will be practiced.
12. Female subjects will need a negative pregnancy screening test if they are of child bearing potential.

Exclusion Criteria:

1. Subjects less than 18 years of age.
2. A lymphocyte doubling time of < 3 months, or other clinical or laboratory signs indicating that a treatment delay of 2 months or longer (due to heavy water labeling and resting period) would result in a significant progression of the disease and be detrimental to the subject, as determined by the treating physician.
3. Any prior treatment for Chronic Lymphocytic Leukemia (CLL) including chemotherapy, chemoimmunotherapy, monoclonal antibody therapy, radiotherapy, or high-dose corticosteroid therapy (Prednisone > 60 mg daily or equivalent), or immunotherapy prior to enrollment or concurrent with this trial.
4. Concomitant use of agents that have been described to affect the biology and/or proliferation rate of CLL cells such as: Phosphodiesterase inhibitors (PDE-inhibitors) (e.g., sildenafil, theophylline), immunosuppressive agents (e.g., prednisone, cyclosporin-A, rapamycin), green tea extract, itraconazole, ketoconazole, clarithromycin, bupropion, and Cox-2 inhibitors.
5. Investigational agent received within 30 days prior to the first dose of study drug. If received any investigational agent prior to this time point, drug-related toxicities must have recovered to Grade 1 or less prior to first dose of study drug.
6. Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
7. Subjects with uncontrolled autoimmune hemolytic anemia (AIHA) or autoimmune thrombocytopenia (ITP).
8. Any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver or other organ system that may place the subject at undue risk to undergo therapy with PCI-32765.
9. Any serious medical condition, laboratory abnormality, or psychiatric illness that places the subject at unacceptable risk if he/she were to participate in the study.
10. History of intracranial hemorrhage or stroke within 6 months prior to the study.
11. Evidence of bleeding diathesis or coagulopathy.
12. Major surgical procedure, open biopsy, or significant traumatic injury, within 28 days prior to Day 1, anticipation of need for major surgical procedure during the course of the study. (Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 1. Bone marrow aspiration +/- biopsy is allowed).
13. Serious, non-healing wound, ulcer, or bone fracture.
14. Subjects receiving anticoagulation (for example heparin, Coumadin, low-molecular-weight heparin (LMWH, such as Lovenox), and anti-platelet drugs (except for low-dose aspirin) will be ineligible to participate in this study. Subjects who recently received drugs for anticoagulation must be off those medications for at least 7 days prior to start of the study.
15. Subjects who are known to be anemic, with hemoglobin <8.0g/dl.
16. Weight less than 110 pounds
17. Subjects who are known to be infected with HIV, or have signs of active Hepatitis B or Hepatitis C.
18. Biliary obstruction, acute hepatitis, severe liver failure, or severely impaired renal function.
19. PCI-32765 is contraindicated in subjects with clinically significant hypersensitivity to any of the compound's structural components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-12-17 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan A. Burger, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kim E, Chen SS, Sivina M, Hwang H, Huang X, Ferrajoli A, Jain N, Wierda WG, Wodarz D, Chiorazzi N, Burger JA. Deuterated water labeling in ibrutinib-treated patients with CLL: leukemia cell kinetics correlate with IGHV, ZAP-70, and MRD. Blood. 2024 Dec 19;144(25):2678-2681. doi: 10.1182/blood.2024025683. PMID 39441901
- [Derived] Burger JA, Li KW, Keating MJ, Sivina M, Amer AM, Garg N, Ferrajoli A, Huang X, Kantarjian H, Wierda WG, O'Brien S, Hellerstein MK, Turner SM, Emson CL, Chen SS, Yan XJ, Wodarz D, Chiorazzi N. Leukemia cell proliferation and death in chronic lymphocytic leukemia patients on therapy with the BTK inhibitor ibrutinib. JCI Insight. 2017 Jan 26;2(2):e89904. doi: 10.1172/jci.insight.89904. PMID 28138560
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 2012 - June 2013
Groups:
- Heavy Water + PCI-32765: 50ml 70% 2^H2O (Heavy Water) 3 times a day for the first 5 days followed by 60 ml daily for a total of 4 weeks (labeling phase). Subjects given first dose in clinic. Subjects then given individual doses of 2^H2O to consume at home; after the 5-day loading period, a 60 ml maintenance dose of 2^H2O will be drunk at bedtime. At end of the 4th week, subjects stop drinking 2^H2O (washout phase) and be followed from 6-12 weeks until beginning treatment with PCI-32765. PCI-32765 administered with 8 ounces (~240mL) of water at a dose of 420 mg (3 x 140mg capsules) orally once daily and continued daily. Treatment duration is 12 cycles, with each cycle consisting of 28 days.
  Heavy Water (2^H2O): 50 ml 70% 2^H2O 3 times a day for the first 5 days followed by 60 ml daily for a total of 4 weeks. After the 5-day loading period, a 60 ml maintenance dose of 2^H2O will be drunk at bedtime. At end of the 4th week, subjects stop drinking 2^H2O (washout phase) and be followed from 6-12
Period: Overall Study
Arm/Group | Heavy Water + PCI-32765
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Heavy Water + PCI-32765
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 64 [48 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Leukemia Cell Death
Description: Stable isotopic labeling with deuterated water (2^H2O) to measure directly the effects of PCI-32765 (ibrutinib) on leukemia cell death in the peripheral blood of participants .
Time Frame: every three months, up to one year
Measure: Median (Full Range); unit: percentage of cell death
Arm/Group | Heavy Water + PCI-32765
Number analyzed (Participants) | 30
percentage of cell death
  Daily death rate of blood cells before therapy | 0.18 [0.0 to 0.7]
  Daily death rate of blood cells after therapy | 1.5 [0.0 to 3.0]

2. Secondary Outcome: Percentage of Recently Born Leukemia Cells Mobilized Into the Blood by PCI-32765 Treatment
Description: Measurement of the fraction of recently born versus older leukemia cells in the peripheral blood of participants before and during PCI-32765 therapy, to determine the effects of PCI-32765 (ibrutinib) therapy on the birth rates of the leukemia cells.
Time Frame: every three months, up to one year
Measure: Median (Full Range); unit: percentage of leukemia cells
Arm/Group | Heavy Water + PCI-32765
Number analyzed (Participants) | 30
percentage of leukemia cells
  Daily cell birth rate before therapy | 0.39 [0.17 to 1.04]
  Daily cell birth rate during therapy | 0.05 [0.0 to 0.36]

ADVERSE EVENTS:
Time Frame: Monthly, for up to 1 year
Arm/Group | Heavy Water + PCI-32765
All-Cause Mortality (participants affected / at risk) | 3/30
Serious Adverse Events (participants affected / at risk) | 16/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heavy Water + PCI-32765 (N=30)
Atrial Fibrillation (Cardiac disorders) | 5 (6)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (2)
Mobitz (tyep)II atrioventricular block (Cardiac disorders) | 1 (1)
Nail Infection (Infections and infestations) | 1 (1)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Pain Extremity (General disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Pleural effusions (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Skin infection (Infections and infestations) | 1 (2)
Suicide attempt (Psychiatric disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heavy Water + PCI-32765 (N=30)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7)
Cardiac Disorders other (Cardiac disorders) | 10 (12)
Gastrointestinal other (Gastrointestinal disorders) | 10 (10)
Hypertension (Vascular disorders) | 9 (9)
Infection (Infections and infestations) | 5 (5)
Oral Mucositis (Gastrointestinal disorders) | 7 (7)
Pain (General disorders) | 23 (26)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 6 (6)
Bruising (General disorders) | 14 (14)
Diarrhea (General disorders) | 16 (16)
Dizziness (Nervous system disorders) | 13 (13)
Dyspena (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Edema (General disorders) | 13 (13)
Fatigue (General disorders) | 21 (21)
Hematuria (Renal and urinary disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin other (Skin and subcutaneous tissue disorders) | 7 (7)
Skin rash (Skin and subcutaneous tissue disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT01752426/Prot_SAP_000.pdf